CLINICAL TRIAL: NCT01582724
Title: Randomized Pragmatic Trial for Women With Menstrual Pain Comparing Additional Self-care Acupressure to Usual Care Alone
Brief Title: Effectiveness of Additional Self-care Acupressure for Women With Menstrual Pain Compared to Usual Care Alone
Acronym: AKUD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Karl and Veronica Carstens Foundation (Other)
Responsible Party: Principal Investigator, Claudia M. Witt, Prof. Dr. med., Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AKUD-12
Record Dates: First submitted 2012-04-18; First posted 2012-04-23 (Estimated); Last update posted 2015-08-04 (Estimated); Status verified 2015-08

CONDITIONS: Menstrual Pain
Keywords: Menstrual pain; Primary dysmenorrhea; Self-care acupressure
MeSH Terms: conditions — Dysmenorrhea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Self-care acupressure (Experimental): 1
  Interventions: Procedure: Self-care acupressure at three predefined points
- Usual care (No Intervention): 2

INTERVENTIONS:
Procedure: Self-care acupressure at three predefined points — Self-care acupressure, one minute for each point, starting 5 days before menstruation, once up to twice daily; when pain is present: twice daily up to five times
  Arms: Self-care acupressure

SUMMARY:
The aim of the study is to evaluate the effectiveness of additional self-care acupressure in women with menstrual pain compared to usual care alone.

DETAILED DESCRIPTION:
Menstrual pain is a common problem in young women and one of the the main reasons of short term absence from school or work. There is some evidence that acupuncture and acupressure might be successful in treating of menstrual pain. Compared with acupuncture, acupressure offers the possibility for women with menstrual pain to do self-care treatment at home. However, studies have been small and self-care acupressure had been only investigated in one study from Taiwan.

ELIGIBILITY:
Inclusion Criteria:

* Women with dysmenorrhea as defined as cramping pain during every menstrual cycle
* Age: 18 to 25 years
* Up to now no prior history of a gynecological disease that could be a reason for dysmenorrhea
* Women with menstruation in the last six weeks and a duration of menstruation cycles between 3 and 6 weeks
* Women with moderate and severe pain defined as a score equal or higher than 6 on the numeric rating scale for the worst pain intensity during the last menstruation.
* Written and oral informed consent
* Women must be able to complete the baseline questionnaire in paper form, the electronic questionnaire via App and a electronic diary via App.
* Presence of a Smartphone and agreement to do data entry through the App

Exclusion Criteria:

* Acupressure, acupuncture, shiatsu- or/and tuina massage at the moment or planned in the next 8 months
* Known or planned pregnancy in the next 8 months.

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 220 (Actual)
Dates: Start 2012-12; Primary Completion 2014-09 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Mean pain intensity at the days of pain during the 3rd cycle after therapy start (Numeric Rating Scale, NRS) | 3rd menstruation after therapy start

SECONDARY OUTCOMES:
Worst pain intensity (NRS) | Baseline, after the 1., 2., 3. and 6. menstruation
Duration of pain | Baseline, after the 1., 2., 3. and 6. menstruation
Responder rate defined as 50% pain reduction at the days of pain | Baseline, after the 1., 2., 3. and 6. menstruation
Sick leave days | Baseline, after the 1., 2., 3. and 6. menstruation
Adverse effects | After 1., 2., 3. and 6. menstruation
Days with medication intake | Baseline, after the 1., 2., 3. and 6. menstruation
Bodily self-efficacy | Baseline, after 1.,2.,3. and 6. menstruation
Credibility of the intervention | After 3. menstruation

CONTACTS AND LOCATIONS:
Overall Officials: Claudia M Witt, MD, Principal Investigator — Institue of Social Science, Epidemiology and Health Economics, Charité University Medical Center Berlin Germany
Locations (1):
- Institue for Social medicine, Epidemiology and Health Economics, Charité University Medical Center, Berlin, Germany

REFERENCES:
- [Derived] Blodt S, Schutzler L, Huang W, Pach D, Brinkhaus B, Hummelsberger J, Kirschbaum B, Kuhlmann K, Lao L, Liang F, Mietzner A, Mittring N, Muller S, Paul A, Pimpao-Niederle C, Roll S, Wu H, Zhu J, Witt CM. Effectiveness of additional self-care acupressure for women with menstrual pain compared to usual care alone: using stakeholder engagement to design a pragmatic randomized trial and study protocol. Trials. 2013 Apr 11;14:99. doi: 10.1186/1745-6215-14-99. PMID 24499425